CLINICAL TRIAL: NCT04895228
Title: Impact of Sacroiliac Joint Injection on Bone Marrow Edema and Disease Outcome Measures in Spondyloarthritis (SpA) Patients
Brief Title: Impact of Sacroiliac Joint Injection on Bone Marrow Edema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sohair Maher mahrous, Sohair Maher Mahrous, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-05-10
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Bone Marrow Edema
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: This study will be a prospective, single-center, randomized, blind clinical trial. It will be performed on patients following in the rheumatology and rehabilitation department in Sohag University Hospitals, Faculty of Medicine:
  N=60 fulfilling ASAS 2010 criteria for axial SpA, will be divided randomly into 2 groups. Group 1 the active group will receive triamcinilone 40 mg injection (Kenacort) + 4 ml of .5 % lidocaine hydrochloride (Xylocaine) under ultrasound guidance. Group 2 will receive similar amount of saline injecteed subcutaneously. Only the patient will be blinded. Particpants will be initially studied with no certain condition for medications wich will be kept unchanged during the study. MRI will be done at base line and BME will be considered as an entry criteria. SPArcc score will be berfoemed at baseline and in the follow-up at 24 weeks post-injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpA patients recieving local steroid injection (Active Comparator): the active group will receive triamcinilone 40 mg injection (Kenacort) + 4 ml of .5 % lidocaine hydrochloride (Xylocaine) under ultrasound guidance.
  Interventions: Procedure: injection
- placebo group (Placebo Comparator): Group 2 will receive similar amount of saline injecteed subcutaneously
  Interventions: Procedure: injection

INTERVENTIONS:
Procedure: injection — triamcinilone 40 mg injection (Kenacort) + 4 ml of .5 % lidocaine hydrochloride (Xylocaine) under ultrasound guidance

SUMMARY:
SpA is a chronic, debilitating inflammatory rheumatic disease that affects axial and peripheral joints, internal organs, and other tissues. Sacroiliitis is a hallmark of axial SpA. Sacroliliitis has a great effect on spine pain, function and cephalic progression of the disease . The prevalence of SpA ranged from 9 to 30 per 10,000 persons in Caucasian populations, Europe or the United States . The management of axial SpA is really challenging. The traditional disease-modifying anti-rheumatic drugs (DMARDs) were ineffective in controlling the axial disease. Biological agents such as tumor necrosis factor alpha (TNFα) inhibitor and anti-interleukin 17 have shown promising results in achieving remission or low disease activity for axial SpA .

Magnetic resonance imaging (MRI) is established as the imaging method of choice for the early diagnosis and follow-up of SpA patients. Although a positive imaging detection of the axial skeleton is no longer obligatory based on the new Assessment of Spondyloarthritis International Society (ASAS) classification criteria 2010, MRI imaging still plays a crucial role, especially in the early diagnosis arm. MRI has a high sensitivity in detection of acute inflammatory processes as well as the high-resolution visualization of anatomical alterations. The lack of radiation exposure makes MRI ideal for monitoring response to treatment .Bone marrow edema (BME) not only showed high sensitivity for detection of early sacroilitis, but also its reduction was a worthy indicator for disease remission. Intra Articular (IA) injections of SIJ with corticosteroids and anesthestics are often performed for pain relief. Although this technique is relatively old, it was not used on a lrage scale in axial SpA patients. Further, its effect on disease outcome measures were not well elucidated. To the best of our knowledge there is no single study have evaluated effect of steroid and local aneshestic injection on improvement of BME . Image guidance of the SIJ injection is fundamanetal, due to the complex anatomy of the joint causing a low accuracy when performed using blind technique .

DETAILED DESCRIPTION:
Study design:

Randomized, double-blinded, prospective, placebo-controlled clinical trial. Aim of the work To evaluate the effectiveness of steroid and anestheisa injection on BME and disease outcome measures in SIJs of axial SpA patients .

Patients and methods

This study will be a prospective, single-center, randomized, blind clinical trial. It will be performed on patients following in the rheumatology and rehabilitation department in Sohag University Hospitals, Faculty of Medicine:

N=60 fulfilling ASAS 2010 criteria for axial SpA, will be divided randomly into 2 groups. Group 1 the active group will receive triamcinilone 40 mg injection (Kenacort) + 4 ml of .5 % lidocaine hydrochloride (Xylocaine) under ultrasound guidance. Group 2 will receive similar amount of saline injecteed subcutaneously. Only the patient will be blinded. Particpants will be initially studied with no certain condition for medications wich will be kept unchanged during the study. MRI will be done at base line and BME will be considered as an entry criteria. SPArcc score will be berfoemed at baseline and in the follow-up at 24 weeks post-injection.

Clinical out come measures including ASDAS BSADAI and BASMI will be performed at baseline and 12 and 24 weeks after SIJ injection.

Inclusion criteria:

* Pateint >18 years old.
* Patients fulfilling ASAS criteria for SpA with a diagnosis confirmed by a rheumatologist.
* Patients having BME of the SIJ on MRI .
* Able to be followed-up regularly.

Exclusion criteria:

* Patient < 18 years old.
* Malignancy, DM, Hepatitis and active infectious disorders
* Spine surgery.
* Ankylosed sacroiliac joint
* Recent SIJ injection

ELIGIBILITY:
Inclusion Criteria:

* Pateint >18 years old.
* Patients fulfilling ASAS criteria for SpA with a diagnosis confirmed by a rheumatologist.
* Patients having BME of the SIJ on MRI .
* Able to be followed-up regularly

Exclusion Criteria:

* Patient < 18 years old.
* Malignancy, DM, Hepatitis and active infectious disorders
* Spine surgery.
* Ankylosed sacroiliac joint
* Recent SIJ injection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
change of bone marrow edema | with in 3 moths
  after steroid injection of sacroiliac joint improvement of bone marrow edema in MRI

CONTACTS AND LOCATIONS:
Overall Officials: sohair maher, Principal Investigator — Sohag University
Locations (1):
- Sohair Maher Mahrous, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No